CLINICAL TRIAL: NCT05150834
Title: Gut Microbiota, the Potential Key to Modulating Humoral Immunogenicity of New Platform COVID-19 Vaccines: Adenovirus-vectored Vaccine Versus mRNA Vaccine
Brief Title: Gut Microbiota, the Potential Key to Modulating Humoral Immunogenicity of New Platform COVID-19 Vaccines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Hye Seong, clinical professor, Korea University Guro Hospital
Other Study IDs: 2021GR0097
Record Dates: First submitted 2021-12-03; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Microbiome; Vaccine; Covid-19; SARS-CoV-2; Immunogenicity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ChAdOx1 vaccinated group: From Febrary 25, 2021 to July 16, 2021, healthy healthcare workers were prospectively recruited at a tertiary hospital in Seoul, Republic of Korea, and they were assigned to get ChAdOx1 (Oxford/AstraZeneca) (n=26) vaccines. Participants were excluded if they had history of medication which would affect gut microbiota in the past 1 month, including antibiotics, laxatives, and motility drugs; previous history of positive SARS-CoV-2 test on nasopharyngeal PCR; or positive serum Spike IgG results.
  Interventions: Other: This is observational study
- BNT162b2 vaccinated group: From Febrary 25, 2021 to July 16, 2021, 53 healthy healthcare workers were prospectively recruited at a tertiary hospital in Seoul, Republic of Korea, and they were assigned to get BNT162b2 (n=27) vaccines. Participants were excluded if they had history of medication which would affect gut microbiota in the past 1 month, including antibiotics, laxatives, and motility drugs; previous history of positive SARS-CoV-2 test on nasopharyngeal PCR; or positive serum Spike IgG results.
  Interventions: Other: This is observational study

INTERVENTIONS:
Other: This is observational study — We enrolled the healthcare workers assigned to get either BNT162b2 or ChAdOx1 by the Korean government.

SUMMARY:
Vaccination is the best way to mitigate the coronavirus disease 2019 (COVID-19) pandemic, but the vaccine immunogenicity may be quite variable from person to person. There is increasing evidence suggesting that the gut microbiome is a major determinant of vaccine immunogenicity. Thus, the investigators investigated the relationship between gut microbiota and humoral immune response after COVID-19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

* People assigned to get either BNT162b2 or ChAdOx1 vaccines
* informed concents

Exclusion Criteria:

* Participants were excluded if they had a history of medication which would affect gut microbiota in the past 1 month, including antibiotics, laxatives, and motility drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From Febrary 25, 2021 to July 16, 2021, 53 healthy healthcare workers were prospectively recruited at a tertiary hospital in Seoul, Republic of Korea, and they were assigned to get either BNT162b2 (n=27) or ChAdOx1 (Oxford/AstraZeneca) (n=26) vaccines. Participants were excluded if they had history of medication which would affect gut microbiota in the past 1 month, including antibiotics, laxatives, and motility drugs; previous history of positive SARS-CoV-2 test on nasopharyngeal PCR; or positive serum Spike IgG results.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Taxonomic biomarkers predicting immune responses | before the administration of first-dose
  This study aimed to analyze whether fecal microbiota composition before vaccination was associated with immmune response level

SECONDARY OUTCOMES:
Antibody titres after the first dose vaccination | 3weeks from the first-dose administration in BNT162b2 group, 8-12weeks from the first-dose administration in ChAdOx1
  This study aimed to analyze maximum immune response after first dose vaccination
Antibody titres after the second dose vaccination | 3 weeks from the second dose administration in both BNT162b2 and ChAdOx1 groups
  This study aimed to analyze maximum immune response after second dose vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Koera University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided